CLINICAL TRIAL: NCT04217395
Title: Implementation and Effectiveness of a Reinforced Support Program for People Who Are Overweight or Obese to Improve Their Autonomy in Health and Quality of Life
Brief Title: Quality of Life and Autonomy in Health of Overweight or Obese People Receiving Reinforced Support
Acronym: Eval-Xailes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: Eval-Xailes_2019
Record Dates: First submitted 2019-12-20; First posted 2020-01-03 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Obesity
Keywords: Obesity; Overweight; Empowerment; Autonomy
MeSH Terms: conditions — Obesity; Overweight; Empowerment | interventions — Adiposity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Reinforced support: X-ailes program users
  Interventions: Behavioral: Obese or overweight health subjects involved in the X-Ailes program (at least one contact with the health system navigator)

INTERVENTIONS:
Behavioral: Obese or overweight health subjects involved in the X-Ailes program (at least one contact with the health system navigator) — The X-Ailes program is a face-to-face or telephone-based support program by health-system navigators and developed by a patients and public association to support overweight or obese care users.
  The main objective of the study is to evaluate the efficacy of the X-ailes program on quality of life of overweight and obese people involved in the program.
  Secondary objectives are to assess their overall health status, their health literacy level and their empowerment. The implementation study is guided by the RE-AIM (Reach, Effectiveness, Adoption, Implementation and Maintenance; Glasgow, Vogt, & Boles, 1999) theoretical framework to determine whether the intervention objectives are being met and to understand the mechanisms of action of the device.

SUMMARY:
This mixed-methods prospective cohort study aims to evaluate a recently implemented reinforced support program named "X-ailes program".

The X-Ailes program is a face-to-face or telephone-based support program by health-system navigators/case-managers, funded by the French Ministry of Health (program for empowerment of care users). X-Ales is developed by an patients and public association to support overweight or obese care users facing difficulty to access to care or resources regarding the management of their health situation.

The subjects of the present study are the overweight or obese care-users followed-up by the X-Ailes program.

The aim of the study Eval-X-ailes is to assess the effect of the support program X-Ailes on quality of life, autonomy and literacy of overweight or obese care users at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18 or more, male or female
* Body mass index equal or over 25
* Resident Living in one of the 2 territories covered by the X-ailes program (Lyon Metropolitan Area or Puy-de-Dôme County)
* Starting Included in the X-ailes program support (1st phone contact to initiate follow-up)
* Not objecting to participating in the evaluation of the X-ailes program

Exclusion Criteria:

* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects are the overweight or obese care health users followed-up byincluded in the X-Ailes program.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2024-05-27 (Estimated); Study Completion 2024-05-27 (Estimated)

PRIMARY OUTCOMES:
Quality of life at 12 months, measured by the specific questionnaire Quality of life, Obesity and Dietetics (QOLOD, Ziegler et al. 2005) | month 12
  The QOLOD questionnaire is adapted to socio-cultural factors of obesity and dietary weight management in France, and it is validated with satisfactory reliability and reproducibility. It contains 36 items grouped into 5 dimensions: physical impact, psycho-social impact, sex-life impact, comfort with food and diet experience. Answers for each question are expressed on a scale from 1 to 5, where 1 =enormously/all the time (true) and 5 = never/not at all (true). Score vary from 0 to 100. Global and dimension scores evolution will measure during the follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- metropolitan area of Lyon, Lyon, France